CLINICAL TRIAL: NCT00838422
Title: Repeatability and Reproducibility of Pachymetric Mapping With Fourier Domain Optical Coherence Tomography, Ocular Response Analyzer, Confoscan 4 and Ultrasound
Brief Title: Reliability of Pachymetry Measurement With FD-oCT, ORA, Confoscan 4 and Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Shu-Wen Chang, Far Eastern Memorial Hospital
Other Study IDs: FEMH97010
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Keratitis
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FD-OCT, ORA, USP

SUMMARY:
The purpose of this study is to assess the repeatability, reproducibility, and agreement of central corneal thickness measured by Fourier Domain Optical Coherence tomography (FD-OCT, OptoVue, USA) with anterior corneal module, 20MHz ultrasound pachymetry equipped with Ocular response analyzer (ORA, Reichert Ophthalmic Instruments, USA) and 10MHz Ultrasound Pachymetry (USP).

DETAILED DESCRIPTION:
Corneal thickness measurements are clinically important. Variation in corneal thickness affects the accuracy of applanation tonometry. A meta-analysis by Doughty and Zaman showed that a 10% change in central corneal thickness may result in an approximately 3.4-mmHg change in intraocular pressure.1 Accuracy of corneal thickness measurement is also important in considering eligibility for refractive surgery, and the amount of correction that can safely be performed. Underestimation of corneal thickness may lead to eligible patients being excluded for primary or enhancement refractive procedures. Overestimation may lead to over-ablation and inadvertent thinning of the stroma, thereby increasing the risk of iatrogenic keratectasia. Hence, studies assessing corneal thickness measurements by various instruments are of high clinical relevance.2-9 Fourier domain optical coherence tomography (FD-OCT, OptoVue, U.S.A), Confoscan 4 (CS-4, Nidek, USA) and ocular response analyzer (ORA, Reichert, USA) are non-invasive medical devices that have recently received FDA approval for measurement of the cornea thickness. However, the repeatability and reproducibility of these instruments remains unproven in the clinical settings. To our knowledge, this is the first study to describe agreement, repeatability and reproducibility in corneal pachymetric mapping between FD-OCT, ORA, CS-4 and conventional ultrasound (US), which has been the current reference corneal pachymetric mapping system for the majority of refractive surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers

Exclusion Criteria:

* Patients who had history of prior ocular surgery, ocular abnormalities other than cataract or refractive error or were unable to cooperate in the examination were excluded.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteer who has no prior ocular disease history and prior intraocular surgical history
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-01 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Repeatability and reproducibility of corneal thickness measurement | 3 months

SECONDARY OUTCOMES:
Comparing central corneal thickness measurement among FD-OCT, ORA, and USP | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Wen Chang, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan